CLINICAL TRIAL: NCT02351999
Title: Clinical Study of the TSP Crosser System For Transseptal Access and Left Atrial Catheter Navigation in Patients Undergoing Atrial Fibrillation Ablation
Brief Title: Clinical Study of the TSP Crosser System for Transseptal Access and Left Atrial Catheter Navigation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Transseptal Solutions Ltd. (Industry)
Collaborators: Meditrial Europe Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CR-14-01
Record Dates: First submitted 2015-01-13; First posted 2015-01-30 (Estimated); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Transseptal puncture; Atrial fibrillation ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TSP Crosser Transseptal Access System (Experimental): The TSP Crosser Transseptal Access System is a novel integrated system combining an extendable radiopaque loop wire to aid in localizing the fossa ovalis (FO); an innovative flexible needle to enable controlled selection of the FO puncture site; and a steerable sheath for enhanced maneuvering and orientation of catheters during LA navigation.
  Interventions: Device: TSP Crosser Transseptal Access System

INTERVENTIONS:
Device: TSP Crosser Transseptal Access System — for transseptal puncture, left atrial access and catheter navigation.

SUMMARY:
The study is a prospective, multi-center, non-randomized single arm interventional investigation with the TSP Crosser Transseptal Access System, a new complete solution for transseptal puncture and left atrial access and catheter navigation, for patients with atrial fibrillation ablation referred for radiofrequency catheter ablation.

DETAILED DESCRIPTION:
Transseptal (TS) catheterization is a critical step for left atrial (LA) interventions (atrial fibrillation ablation, LA appendage closure, mitral valve interventions). The availability of suitable tools and techniques is essential to safely perform the TS puncture, effectively deliver radiofrequency lesions, deploy LA devices, and anticipate difficult procedural situations in which complications may arise. This study is intended to assess the safety, performance and usability of the TSP Crosser System in facilitating access to the left atrium and catheter navigation to the pulmonary veins (PV) during catheter based ablation procedures for the treatment of atrial fibrillation (AF). Moreover, the study will assess the impact of the TSP Crosser System on procedural times, including time to achieve left atrial accesses, total procedure times, total fluoroscopy time, left atrial mapping time and radiofrequency isolation times. The study is a prospective, multicenter, non-randomized single arm interventional investigation. Enrolled subjects who meet the study inclusion/exclusion criteria will be evaluated during the catheter mapping and ablation procedures and followed until release from hospital post procedure per institutional standard of care. After 30 days, patient will be contacted by telephone to obtain information on their clinical condition and any adverse events; if necessary, a clinic visit may be performed when required by the physician.

ELIGIBILITY:
Inclusion Criteria:

* Patient is referred to receive a catheter ablation procedure for atrial fibrillation, requiring transseptal access and LA catheterization
* Patient has signed the informed consent form and is willing to participate in the clinical study and data collection
* Patient age is between 18 and 80 years old

Exclusion Criteria (Procedure Related): The use of the TSP Crosser System is contraindicated in patients with the following conditions:

* Atrial thrombus or tumor or myxoma.
* Previous interatrial septal patch or prosthetic atrial septal defect closure device.
* Interruption of inferior vena cava.
* Giant right atrium (70 mm diameter or more).
* Severe rotational anomalies of the heart or great vessels
* Severe kyphoscoliosis.
* Marked dilation of the ascending aorta.
* Inability to lie flat.

Exclusion Criteria (Clinical): Subjects with following conditions will also be considered unsuitable for enrollment:

* Unstable angina or ongoing myocardial infarction.
* History of recent systemic arterial embolization (within 1 month).
* History of recent Cerebral Vascular Accident (CVA) (within 1 month).
* Active infection or sepsis.
* Enrollment in any other ongoing study protocol.
* Female patient is pregnant or lactating.
* Untreatable allergy to contrast media or device materials in contact with blood or skin (Pebax, PTFE, Nitinol, Stainless steel, Polycarbonate, ABS, silicon, acetal, Pet-P (Ertalyte), POM (Delerin), Polycarbonate).
* Unable to tolerate anticoagulation therapy (heparin or warfarin).
* History of blood clotting (bleeding or thrombotic) abnormalities, with increased risk of bleeding.
* Any other health condition that, in the opinion of the investigator, makes the subject unsuitable for transseptal left atrial catheterization
* Participation in concomitant research studies of investigational products.
* Subject will not agree to return to the implant center for the required number of follow-up visits or is geographically unavailable for follow-up.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-06-15 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Ability to achieve transseptal access | intraoperative
  Ability to achieve transseptal access with the TSP Crosser needle with the aid of the loopwire for locating the fossa ovalis. The ability to achieve transseptal access will be assess by the successful puncture of the TSP Crosser needle and by the utility of TSP Crosser loop wire for locating the fossa ovalis (graded by the investigators with a Likert scale: from 1 = unacceptable to 5 = excellent, unit value)
TSP Crosser Introducer steerability and positioning for ablation catheter placement | intraoperative
  TSP Crosser Introducer steerability and positioning to facilitate ablation catheter placement as seen fluoroscopically and by ability to visualize navigation of ablation catheter to the pulmonary veins. Outcome will be assessed by ability of ablation catheter to be inserted and retrieved through the sheath visualized fluoroscopically during the procedure, graded by the investigators with a Likert scale (from 1 = unacceptable to 5 = excellent, unit value)
TSP Crosser System usability | intraoperative
  TSP Crosser System usability, graded by the investigators with a Likert scale (from 1 = unacceptable to 5 = excellent, unit value)

SECONDARY OUTCOMES:
Overall serious adverse events (SAE)/complication rate (in percentage). Complications will be analyzed and grouped as device-related, procedure-related and other complications. | at the end of procedure; up to 10 days from index treatment; at 30 days after index treatment
Duration of Procedural Endpoints | intraoperative
  * Evaluation of the time to achieve left atrial access (in minutes)
  * Total procedural time (in minutes)
  * Total fluoroscopy time (in minutes)
  * Left atrial mapping time (in minutes)
  * Radiofrequency pulmonary veins isolation time (in minutes).

CONTACTS AND LOCATIONS:
Overall Officials: Monica Tocchi, MD, PhD, Study Director — Meditrial Europe Ltd.
Locations (2):
- CHU Bichat-Claude Bernard, Paris, France
- Asklepios Klinik St. Georg, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided